CLINICAL TRIAL: NCT02540811
Title: A Prospective, Non-comparative Clinical Investigation of a Novel Decellularised Porcine Xenograft (dCELL® ACL Scaffold) for Reconstruction of the Anterior Cruciate Ligament
Brief Title: Clinical Evaluation of dCELL® ACL Scaffold for Reconstruction of the Anterior Cruciate Ligament
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tissue Regenix Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRG-A01-01
Record Dates: First submitted 2015-08-26; First posted 2015-09-04 (Estimated); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Knee Injuries
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dCELL® ACL Scaffold (Experimental)
  Interventions: Device: dCELL® ACL Scaffold

INTERVENTIONS:
Device: dCELL® ACL Scaffold

SUMMARY:
The safety and performance of dCELL® ACL Scaffold will be evaluated in 40 patients who have been implanted with the investigational product following a ruptured anterior cruciate ligament (ACL) of the knee.

DETAILED DESCRIPTION:
The dCELL® ACL Scaffold is a novel device manufactured from porcine tissue using a patented variation of Tissue Regenix's platform technology to render the tissue biocompatible and free from cellular material, providing a biological scaffold that is safe for human implantation whilst preserving the biomechanical properties.

The device is used to reconstruct traumatic ACL tears to help restore normal knee function and therefore prevent further wear of the cartilage and future damage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with partial or complete tear of the ACL and require reconstruction of the ACL.
* Medial Collateral Ligament (MCL) injury grade 2 or less.
* Osteoarthritis grade 2 or less on the Kellgren Lawrence scale.
* Patients who have given written informed consent; and are willing and able to comply with entire study procedures including rehabilitation protocol.

Exclusion Criteria:

* Body Mass Index (BMI) greater than 35 kg/m2.
* Treatment with any investigational drug or device within two months prior to screening.
* Patients presenting with abnormal degenerative osteoarthritis of the joint.
* Previous ACL reconstruction on the target knee.
* Current ACL injury on contralateral knee.
* Patients using anticoagulants within 2 weeks prior to surgery.
* Patients on current immuno-suppressive or radiation therapy within six months of screening.
* Patients with diabetes or cardiovascular disease which precludes elective surgery.
* Patients with documented renal disease or metabolic bone disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2021-08-11 (Actual); Study Completion 2021-08-11 (Actual)

PRIMARY OUTCOMES:
Arthrometric measurement of knee joint laxity | Baseline, 3 months, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Comparison of the magnitude of side-to-side differences in mm between the treated knee and the opposite normal knee using an arthrometric ligament testing device
Lachman Test | Baseline, 3 months, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Clinical assessment of knee stability
Pivot Shift Test | Baseline, 3 months, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Clinical assessment of knee stability
Number of Participants With Treatment-Related Adverse Events | Surgery, 3 months, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  The frequency and seriousness of any adverse events or adverse device effects will be assessed

SECONDARY OUTCOMES:
Outcome measure questionnaire of knee functional improvement in terms of symptoms, sport activities and ability to function | Baseline, 3 months, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Patient's subjective score of 1 to 100 points, with 100 implying the best results and 1 the worst results
Evidence of integration of the investigational product by MRI | Baseline, 3 months, 6 months, 12 months, 24 months
  Changes to the articular cartilage or joint space at follow up time points compared to pre-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Simon Roberts, Principal Investigator — The Robert Jones & Agnes Hunt Orthopaedic Hospital NHS Foundation Trust
Locations (8):
- Poland (2):
  - Klinika Chirurgii Endoskopowej Sp. z o.o., Żory, Ul. Bankowa 2
  - Med-Polonia Sp. z o.o., Poznan, Ul. Obornicka 262
- Spain (4):
  - Hospital Infanta Elena de Madrid-Valdemoro, Madrid, Avd. Reyes Catolicos, 21
  - Hospital Clinico San Carlos, Madrid, Calle Profesor Martin Lagos
  - Hospital Universitario La Ribera de Alzira, Valencia, Carretera Corbera, Km1
  - Hospital Universitari de Bellvitage, Barcelona, L'Hospilatet de Llobregat
- United Kingdom (2):
  - Clifton Park Hospital, York, North Yorkshire
  - Robert Jones and Agnes Hunt Hospital NHS Foundation Trust, Oswestry, Shropshire